CLINICAL TRIAL: NCT06918886
Title: Evaluation of Liver Fibrosis and Hepatic Steatosis Using FIB-4 Score and Ultrasonography in Psoriatic Arthritis Patients Treated With TNF or IL-17 Inhibitors: A Retrospective Controlled Study
Brief Title: Comparison of Liver Health in Psoriatic Arthritis Patients Using Anti-TNF or Anti-IL17 Treatments
Acronym: FIB-4 PsA
Status: Not yet recruiting | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/400
Record Dates: First submitted 2025-03-17; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Psoriatic Arthritis (PsA); Liver Fibrosis; Liver Diseases
Keywords: Psoriatic Arthritis; Liver Fibrosis; FIB-4 Score; Anti-TNF Therapy; Anti-IL17 Therapy; Biological Therapy; Liver Health; Retrospective Study; Hepatic Safety; Chronic Inflammatory Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Liver Cirrhosis; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Anti-TNF treatment: Psoriatic arthritis patients with outcome assessment at 24 months following the initiation of Anti-TNF biological treatment.
- Group 2: Anti-IL17 treatment: Psoriatic arthritis patients with outcome assessment at 24 months following the initiation of Anti-IL-17 biological treatment.
- MTX Control Group: This cohort comprises psoriatic arthritis (PsA) patients with outcome assessment at 24 months following the initiation of methotrexate (MTX) monotherapy. They will serve as the control group to compare the effects on liver health with those treated using biologic agents. No other specific interventions beyond standard MTX therapy are administered to this group.

SUMMARY:
Psoriatic arthritis (PsA) is an inflammatory joint disease that can also affect the liver. Some medications used to treat PsA, such as biological agents (TNF-alpha inhibitors and IL-17 inhibitors), may influence liver health over the long term. This retrospective study aims to evaluate the presence and progression of liver fibrosis (scarring) and hepatic steatosis (fatty liver) in PsA patients treated with TNF-alpha inhibitors or IL-17 inhibitors.

The study includes PsA patients who have used biological medications continuously for at least 2 years. Patients' liver health will be assessed using non-invasive tests such as liver ultrasonography and validated biochemical scoring systems (FIB-4, APRI). The findings will be compared with PsA patients treated only with methotrexate (MTX), a commonly used medication known to affect liver health.

This study will help understand whether biological therapies (TNF or IL-17 inhibitors) have a positive or negative impact on liver health compared to traditional treatments (MTX) in patients with psoriatic arthritis.

DETAILED DESCRIPTION:
This is a retrospective, single-center observational study, conducted in the Physical Medicine and Rehabilitation Clinic, designed to assess the impact of long-term biologic therapy on liver health in patients with psoriatic arthritis (PsA). Participants must have received either TNF-alpha inhibitors or IL-17 inhibitors for at least two consecutive years. A separate group of PsA patients who have only received methotrexate (MTX) for at least two years will serve as a comparison cohort.

Objectives:

To estimate the frequency of hepatic steatosis and fibrosis using liver ultrasonography and validated biochemical scoring indices (FIB-4, APRI) among patients on biologic therapy and MTX.

To compare changes in fibrotic markers between baseline and the two-year follow-up period.

To determine whether long-term biologic therapy poses additional risk or provides any protective effect regarding the progression of liver disease.

Study Population:

Adult PsA patients aged 18 to 65 years, meeting standard classification criteria.

Biologic therapy group: ongoing anti-TNF or anti-IL-17 treatment for ≥2 years.

Control group: MTX therapy ≥2 years without biologic agents.

Methods:

Patient records from the rheumatology department will be reviewed retrospectively.

Liver ultrasonography, performed at baseline (or earliest available pre-biologic record) and at the two-year mark, will evaluate hepatic steatosis, if available in patient files.

Blood tests (AST, ALT, platelet count, total bilirubin, albumin, CRP) will be retrieved from clinical databases to calculate non-invasive liver fibrosis indices (e.g., FIB-4, APRI). Additional data on metabolic risk factors (BMI, diabetes, hypertension, dyslipidemia measured by total cholesterol, LDL, HDL, and triglyceride levels) will be extracted. Additionally, clinical information on enthesitis, dactylitis, and disease activity (assessed by DAPSA and/or PASI scores when available) will be recorded from patient files.

Statistical analysis will include group comparisons, correlation analyses, and multiple regression to adjust for confounding factors.

Significance:

Findings from this study will enhance understanding of whether TNF-alpha or IL-17 inhibitors elevate or mitigate the risk of liver disease progression relative to MTX therapy in PsA patients, providing a foundation for more tailored treatment decisions and long-term patient monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years
* Diagnosed with psoriatic arthritis (PsA) according to standard classification criteria
* Receiving biologic therapy (anti-TNF or anti-IL-17) or MTX monotherapy for ≥2 years
* Able to provide historical data (medical records) on liver ultrasound and laboratory parameters

Exclusion Criteria:

* History of any other chronic liver disease (e.g., viral hepatitis, autoimmune hepatitis)
* Significant alcohol consumption (>20 g/day women, >30 g/day men)
* Concomitant use of other hepatotoxic drugs apart from MTX
* Unwillingness or inability to comply with study assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study population comprises adult PsA patients (aged 18 to 65) under active follow-up at the Physical Medicine and Rehabilitation Clinic. Eligible participants have confirmed PsA diagnoses and must have been treated either with methotrexate (MTX) alone or with biologic agents (anti-TNF or anti-IL-17) for at least two years. Data from medical records-including liver ultrasound reports, laboratory results, and relevant clinical assessments-will be collected retrospectively. Patients with significant alcohol use or other known causes of chronic liver disease are excluded. The sample is expected to encompass a range of disease severities, allowing for meaningful comparison of liver health outcomes across different therapeutic regimens.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Liver Health using Fibrosis-4 (FIB-4) Index Score | Outcome assessment at 24 months post-treatment initiation
  The Fibrosis-4 (FIB-4) Index is a tool used for the noninvasive assessment of liver fibrosis. Comparison of liver fibrosis scores (FIB-4) calculated from AST, ALT, platelet counts, and age between Anti-TNF and Anti-IL17 treated Psoriatic Arthritis patients. There is no fixed minimum or maximum value; however, the following threshold values are commonly used in clinical interpretation:
  <1.3: Low likelihood of advanced fibrosis 1.3-2.67: Indeterminate/intermediate risk >2.67: High likelihood of advanced fibrosis. Higher FIB-4 scores indicate the presence of more advanced liver fibrosis.

SECONDARY OUTCOMES:
Identification of High-Risk Patients | Outcome assessment at 24 months post-treatment initiation
  Determining the percentage of patients with elevated FIB-4 scores suggestive of liver fibrosis risk in each treatment group (Anti-TNF vs. Anti-IL17).Higher FIB-4 scores indicate the presence of more advanced liver fibrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Serkan Kılıçoğlu, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient confidentiality concerns and the retrospective nature of the data collection, which may limit consent for data sharing.

REFERENCES:
- [Background] Verhoeven F, Weil-Verhoeven D, Prati C, Martino VD, Thevenot T, Wendling D. Safety of TNF inhibitors in rheumatic disease in case of NAFLD and cirrhosis. Semin Arthritis Rheum. 2020 Aug;50(4):544-548. doi: 10.1016/j.semarthrit.2020.03.013. Epub 2020 May 11. PMID 32446022
- [Background] Verhoeven F, Prati C, Di Martino V, Thevenot T, Demougeot C, Wendling D, Weil-Verhoeven D. Evolution of FIB-4 score in SpA and PsA patients taking anti-TNF or anti-IL17. Joint Bone Spine. 2024 Dec;91(6):105763. doi: 10.1016/j.jbspin.2024.105763. Epub 2024 Jul 29. No abstract available. PMID 39084400